CLINICAL TRIAL: NCT03023332
Title: Tailored Health Self-Management Interventions for Highly Distressed Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jaclene A. Zauszniewski, Principal Investigator, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01NR016817-01 (NIH)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Distress; Caregiver
Keywords: Caregiver; Biofeedback; Resourcefulness; Self-Management

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-management need (Experimental): SM-need (i.e. need for bipolar education or resourcefulness training or HRV-focused biofeedback training or no need for any)
  Interventions: Behavioral: Resourcefulness Training; Behavioral: Biofeedback training; Behavioral: Bipolar Education
- Self-management preference (Experimental): SM-preference (i.e. preference for bipolar education or resourcefulness training or HRV-focused biofeedback training or no intervention)
  Interventions: Behavioral: Resourcefulness Training; Behavioral: Biofeedback training; Behavioral: Bipolar Education
- Control (No Intervention): No intervention or treatment
- Usual care (Active Comparator): Bipolar education
  Interventions: Behavioral: Bipolar Education

INTERVENTIONS:
Behavioral: Resourcefulness Training — A cognitive-behavioral intervention delivered through iPad technology that consists of teaching and reinforcing personal (self-help) and social (help-seeking) resourcefulness skills.
  Arms: Self-management need; Self-management preference
Behavioral: Biofeedback training — Use of a heart-rate variability (HRV) tracking device to enable one to learn to alter physiology to improve health. Devices are used to measure physiological activity, e.g., breathing and heart function, and provide rapid, accurate "feedback" to the user, thereby enabling desired physiological changes that can endure over time without continued use of the device and continue to influence behavior.
  Arms: Self-management need; Self-management preference
Behavioral: Bipolar Education — An educational program designed to teach family caregivers of about the types, causes, symptoms, episodes, warning signs, and treatments for individuals with bipolar disorder, as well as available resources for assisting a family member with bipolar disorder. The content to be presented within an audiovisual format using iPad technology follows the recommendations and guidelines developed through research and by the Depression and Bipolar Support Alliance and the National Institute of Mental Health.
  Arms: Self-management need; Self-management preference; Usual care

SUMMARY:
How do varying levels of participation in selecting self-management interventions (ranging from no input into the selection to selection based on need or preference) affect health risks and physical and mental health over time in family caregivers of persons with bipolar disorder? Caregivers will be randomized to: 1) a control group (no intervention); 2) education (usual care); 3) self-management intervention based on need (SM-need); or 4) self-management intervention of their preference (SM-preference).

DETAILED DESCRIPTION:
The study has two aims: The primary aim (A1) is to examine differences across the four groups (control, usual care, SM-need, and SM-preference) on caregiver health (health risks and mental and physical health) over time. We hypothesize that the caregivers who receive a self-management intervention based on need (SM-need) or preference (SM-preference) will have better health outcomes than those in the usual care or control groups.

Secondary aims are to: A2) explore whether caregiver baseline need or preference for intervention (i.e. choice) is associated with: a) care recipient's symptoms; b) caregiver reactions; and c) caregiving involvement, and A3) build caregiver profiles from demographic/ contextual factors that are associated with their needs and preferences for the self-management interventions.

All caregivers will complete assessment measures and measures of health risks, and physical and mental health at baseline (T1), 6 months (T2) and 12 months (T3). Caregivers will randomly assigned to one of four groups. The control group will receive no intervention. The usual care group will receive bipolar education. The SM-need group will receive a self-management intervention tailored to meet their need for bipolar education, biofeedback training, or resourcefulness training, as determined by baseline cut scores. Caregivers in the SM-preference group will choose one of the three self-management intervention according to their personal preference.

All three self-management interventions (bipolar education, biofeedback training, resourcefulness training) are delivered over four weeks (between T1 and T2). Caregivers may use the one SM intervention whenever and as often as they wish (i.e. self-tailoring) for the remainder of the study period. The bipolar education and resourcefulness training interventions will be delivered initially using an iPad. These interventions involve providing educational information about bipolar disorder or teaching self-help (stress-management, problem-solving) and help-seeking skills, respectively. Biofeedback training consists of use of a hand-held device that shows the participant their changes in heart rate based on changes in their breathing pattern (as they relax); caregivers who need or prefer the biofeedback will be given a device to use for 28 days. All study participants receiving the intervention will also be asked to keep a journal to record their experience with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* At least 18 years old
* Have a family member with bipolar disorder
* Have cared/supported them for at least the last 6 months in the last year
* Be capable of performing the informed consent and participate in interventions

Exclusion Criteria:

* Does not have family member with bipolar disorder
* Has not cared for family member for at least 6 months in the last year
* Knowledge of another family member in the same household enrolled in the study
* Is pregnant
* Has a pacemaker
* Lives outside of the study area (Cuyahoga, Lake, Geauga, Portage, Summit, Medina, and Lorain counties)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclene Zauszniewski, PhD, Principal Investigator — Case Western Reserve University - Frances Payne Bolton School of Nursing
Locations (1):
- CWRU School of Nursing, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zauszniewski JA, Burant CJ, Juratovac E, Jeanblanc A, Sweetko JS, Larsen C, Almutairi R, She HY, DiFranco E, Colon-Zimmerman K, Sajatovic M. Acquiring Resourcefulness Skills: Formal Versus Informal Training. West J Nurs Res. 2025 Jan;47(1):5-14. doi: 10.1177/01939459241296613. Epub 2024 Nov 13. PMID 39535112

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The only participants excluded from assignment signed a consent form but withdrew or did not respond to requests to complete T1. We do not report their subdivision into self-management interventions as, per our study Aims, we were not looking at the effects of the individual self-management interventions.
Period: Overall Study
Arm/Group | Self-management Need | Self-management Preference | Control | Usual Care
Started | 86 | 86 | 70 | 68
Completed | 62 | 65 | 58 | 48
Not Completed | 24 | 21 | 12 | 20
Not completed — Withdrawal by Subject | 10 | 5 | 4 | 7
Not completed — Lost to Follow-up | 13 | 16 | 8 | 13
Not completed — Death | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the baseline T1 questionnaire
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-management Need | Self-management Preference | Control | Usual Care | Total
Number analyzed (Participants) | 86 | 86 | 70 | 68 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 73 | 73 | 60 | 59 | 265
  >=65 years | 13 | 13 | 10 | 9 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.24 (13.98) | 51.14 (14.39) | 51.64 (13.46) | 49.4 (14.65) | 50.98 (14.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 66 | 53 | 52 | 235
  Male | 22 | 20 | 17 | 16 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 37 | 27 | 24 | 29 | 117
  White | 46 | 49 | 39 | 38 | 172
  More than one race | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 2 | 7 | 5 | 1 | 15
Region of Enrollment [Number; unit: participants]
  United States | 86 | 86 | 70 | 68 | 310
Resourcefulness [Mean (Standard Deviation); unit: units on a scale] — Resourcefulness scale score. Composite item comprising of responses to 28 items scored on a 6 point likert scale. Scores range from 0-140, with higher scores indicating greater resourcefulness.
  units on a scale | 90.05 (18.14) | 91.10 (13.38) | 91.26 (19.15) | 94.78 (18.31) | 93.38 (17.64)
Bipolar knowledge score [Mean (Standard Deviation); unit: units on a scale] — The scale measures caregiver knowledge of bipolar disorder using a 16 item scale. Scores range from 0-43, with higher scores indicating greater knowledge.
  units on a scale | 21.94 (3.36) | 22.08 (3.55) | 22.16 (3.55) | 21.59 (3.39) | 22.05 (3.49)
Health Risks [Mean (Standard Deviation); unit: units on a scale] — Health risks were measured using the Change in Health Risk Behavior Scale. The scale consists of 9 items measured on a 3-point scale, Scores range 9-27; higher score indicates greater risk
  units on a scale | 15.77 (2.94) | 14.98 (2.89) | 15.13 (2.89) | 15.01 (2.67) | 15.24 (2.86)
Global Health [Mean (Standard Deviation); unit: units on a scale] — Change in Global Health - PROMIS (Patient Reported Outcomes Measurement Information System) scale. 5 items - physical health; 5 items - mental health; 5-point scale; Scores range 0-40; higher scores indicate better health.
  units on a scale | 25.59 (5.43) | 27.28 (4.89) | 26.657 (4.79) | 26.43 (5.49) | 26.47 (5.16)

OUTCOME MEASURES:

1. Primary Outcome: Change in Caregiver Health - Health Risks
Description: Health risks were measured using the Change in Health Risk Behavior Scale. The scale consists of 9 items measured on a 3-point scale, Scores range 9-27; higher score indicates greater risk
Time Frame: 12 months
Population: All participants completing T1 and T3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-management Need | Self-management Preference | Control | Usual Care
Number analyzed (Participants) | 59 | 60 | 53 | 48
score on a scale
  T1: Baseline | 15.53 (2.96) | 14.65 (2.85) | 15.02 (2.79) | 14.80 (2.91)
  T3: 12 month followup | 14.84 (3.31) | 15.00 (3.12) | 14.91 (2.86) | 15.16 (3.99)

2. Primary Outcome: Change in Global Health - PROMIS (Patient Reported Outcomes Measurement Information System)
Description: Change in Global Health - PROMIS (Patient Reported Outcomes Measurement Information System) scale. 5 items - physical health; 5 items - mental health; 5-point scale; Scores range 0-40; higher scores indicate better health.
Time Frame: 12 months
Population: All participants completing T1 and T3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-management Need | Self-management Preference | Control | Usual Care
Number analyzed (Participants) | 59 | 84 | 53 | 48
score on a scale
  T1: Baseline | 25.95 (5.27) | 27.77 (4.99) | 26.66 (4.61) | 27.54 (5.37)
  T3: 12 month followup | 27.45 (4.97) | 27.4 (5.95) | 26.62 (5.46) | 28.42 (5.27)

3. Secondary Outcome: Change in Bipolar Knowledge Assessment Scale
Description: The scale measures caregiver knowledge of bipolar disorder using a 16 item scale. Scores range from 0-43, with higher scores indicating greater knowledge.
Time Frame: 12 months
Population: All participants completing both T1 and T3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-management Need | Self-management Preference | Control | Usual Care
Number analyzed (Participants) | 59 | 60 | 53 | 48
score on a scale
  T1: Baseline | 21.90 (3.62) | 22.58 (3.31) | 22.11 (3.64) | 21.48 (3.37)
  T3: 12 month followup | 22.29 (3.55) | 21.85 (3.75) | 22.47 (3.69) | 21.69 (3.54)

4. Secondary Outcome: Change in Heart Rate Variability
Description: HRV is a physiological measure of the healthy functioning of the heart. It is a well-established biomarker for detecting stress. HRV was measured using the BioRadio portable limb-lead electrocardiogram recorder. A sensor was placed on the radial area of the caregiver's forearm for 5 minutes; they were asked to remain still as possible to prevent artifacts in the readings. The data obtained via this device was analyzed with compatible VivoSense software, which automatically computed 8 HRV parameters. One of these was the SDNN score, which is the recognized and most commonly used gold standard biomarker indicative of stress. The SDNN score is the standard deviation of all normal to normal R-R intervals between heartbeats and reported in milliseconds. The SDNN was the outcome of interest for our study as a physiological indicator of stress. For each caregiver, the software produced an average score for the 5-minute measurement
Time Frame: 12 months
Population: Participants completing both T1 and T3 questionnaires.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Self-management Need | Self-management Preference | Control | Usual Care
Number analyzed (Participants) | 59 | 60 | 53 | 48
milliseconds
  T1: Baseline | 56.64 (57.82) | 50.41 (30.57) | 67.94 (147.48) | 57.07 (36.18)
  T3: 12 month followup | 63.34 (50.67) | 59.53 (35.67) | 69.58 (76.63) | 44.14 (28.85)

5. Secondary Outcome: Change in Resourcefulness
Description: Participant Resourcefulness scale score. Composite item comprising of responses to 28 items scored on a 6 point likert scale. Scores range from 0-140, with higher scores indicating greater resourcefulness.
Time Frame: 12 months
Population: All participants completing T1 and T3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-management Need | Self-management Preference | Control | Usual Care
Number analyzed (Participants) | 59 | 60 | 53 | 48
score on a scale
  T1: Baseline | 92.93 (17.29) | 92.78 (13.79) | 93.15 (20.1) | 94.83 (19.72)
  T3: 12 month followup | 92.82 (19.37) | 93.81 (15.87) | 94.29 (19.24) | 96.49 (17.88)

ADVERSE EVENTS:
Time Frame: Data was collected for the duration of the study. Participants completed a baseline questionnaire (T1), a 1 month intervention, and followup questionnaires at 6months (Q2) and 12 months (Q3) post-intervention.
Arm/Group | Self-management Need | Self-management Preference | Control | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/86 | 0/86 | 0/70 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86 | 0/70 | 0/68
Other Adverse Events (participants affected / at risk) | 0/86 | 0/86 | 0/70 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT03023332/Prot_SAP_000.pdf